CLINICAL TRIAL: NCT05348265
Title: Effects of High Intensity Interval Training on Psychological Well Being, Anthropometrics, and Quality of Life in Females With Polycystic Ovarian Syndrome
Brief Title: High Intensity Interval Training in PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SanaRasheed
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Intensity steady state training (Active Comparator): Intervention will be provided for a period of 8 weeks. For the first 4 weeks the intervention will consist of 35-40 minutes of supervised slow paced treadmill walk, five days a week. From week 5 till 8 the intervention will consist of 50-60 minutes of supervised slow paced treadmill walk, five days a week.
  Interventions: Other: Low Intensity steady state training
- High intensity interval training (Experimental): Intervention will be provided for a period of 8 weeks, thrice a week. Intervention will start with a 5 minutes warm up period of jogging in place. For the first 4 weeks, 3 series of these exercises will be performed with 3 minutes of rest in between: 30 seconds burpees + 30 seconds recovery, 30 seconds lunges + 30 seconds recovery, 30 seconds skipping + 30 seconds recovery, 30 seconds squats + 30 seconds recovery.
  Exercise session will be followed by a cool down of 5 to 10 minutes with upper and lower extremity stretches.
  Intervention will start with a 5 minutes warm up period of jogging in place. For weeks 5 to 8, 4 series of these exercises will be performed with 3 minutes of rest in between: 30 seconds burpees + 30 seconds recovery, 30 seconds lunges + 30 seconds recovery, 30 seconds skipping + 30 seconds recovery, 30 seconds squats + 30 seconds recovery.
  Exercise session will be followed by a cool down of 5 to 10 minutes with upper and lower extremity stretches.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: Low Intensity steady state training — Intervention will be provided for a period of 8 weeks. For the first 4 weeks the intervention will consist of 35-40 minutes of supervised slow paced treadmill walk, five days a week. From week 5 till 8 the intervention will consist of 50-60 minutes of supervised slow paced treadmill walk, five days a week.
  Arms: Low Intensity steady state training
Other: High intensity interval training — Intervention will be provided for a period of 8 weeks, thrice a week. Intervention will start with a 5 minutes warm up period of jogging in place. For the first 4 weeks, 3 series of these exercises will be performed with 3 minutes of rest in between: 30 seconds burpees + 30 seconds recovery, 30 seconds lunges + 30 seconds recovery, 30 seconds skipping + 30 seconds recovery, 30 seconds squats + 30 seconds recovery.
  Exercise session will be followed by a cool down of 5 to 10 minutes with upper and lower extremity stretches.
  Intervention will start with a 5 minutes warm up period of jogging in place. For weeks 5 to 8, 4 series of these exercises will be performed with 3 minutes of rest in between: 30 seconds burpees + 30 seconds recovery, 30 seconds lunges + 30 seconds recovery, 30 seconds skipping + 30 seconds recovery, 30 seconds squats + 30 seconds recovery.
  Exercise session will be followed by a cool down of 5 to 10 minutes with upper and lower extremity stretches.
  Arms: High intensity interval training

SUMMARY:
Study objective is to determine the effect of High intensity interval training on psychological wellbeing, Anthropometrics and Quality of life in females with Polycystic Ovarian Syndrome

ELIGIBILITY:
Inclusion Criteria:

* females 18 to 45 years of age
* Diagnosed with PCOS based on Rotterdam criteria
* Ferriman and Gallway score of >8 for hirsutism

Exclusion Criteria:

* Use of hormonal contraceptives or IUDs for contraception
* Taking metformin <3 months prior to the inclusion
* Breast feeding mothers
* Type I or II DM
* Hypo/hyperthyroidism
* Regular high-intensity endurance or strength training (defined as ≥ 2 sessions of vigorous exercise per week), Physical ailments/injuries that limited exercise performance.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Mental Well-being | 8th Week
  Changes from the baseline Warwick Edinburgh Mental Well-being Scale is a 14 item scale of mental well-being covering subjective well-being and psychological functioning, in which all items are worded positively and address aspects of positive mental health. The scale is scored by summing responses to each item answered on a1 to5 scale. The minimum scale score is 14 and the maximum is 70.
Illness perception | 8th Week
  Changes from the baseline The Brief Illness Perception Questionnaire (IPQ) it consists of 9 items rated on a scale of 0 to 10. First five items asses such as effect on life (item 1); duration of illness (item 2); control over illness (item 3); beliefs about the effectiveness of treatment (item 4); and experience of symptoms (item 5). Items 6 and 8 assess emotional aspects to include concern about illness and a multifaceted question about mood. Item 7 assesses degree of understanding of the illness. The final item is open-ended, asking respondents to rank the three most important factors causing their illness. . A higher score reflects a more threatening view of the illness.
weight | 8th week
  Changes from the baseline the Weight will be measured using a digital weighing scale in kilograms.
BMI | 8th week
  Changes from the baseline the BMI will be measured by dividing weight in kilograms by height in centimeters. BMI Asian will be used for categorization i.e. less than 18.5 kg/m2 is underweight, 18.5 to 23 18.5 kg/m2 is normal, 23 to 27.5 18.5 kg/m2 is overweight and more than 27 18.5 kg/m2 is obese.
waist-to-hip ratio | 8th Week
  changes from the baseline waist to hip ratio will be measured using a measuring tape. A score of less than 0.8 is considered normal, 0.81 to 0.85 is moderate and more than 0.86 is higher.

SECONDARY OUTCOMES:
Polycystic ovary syndrome health-related Quality of life questionnaire | 8th Week
  Changes from the baseline The PCOSQ contains the following domains: emotions (8 items), hirsutism (5 items), weight (5 items), infertility (4 items), and menstrual disorders (4 items). Each item can be answered by choosing from a Likert scale with 7 options from 1 (always) to 7 (never). Higher scores are indicative of better function.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ehsan, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No